CLINICAL TRIAL: NCT04266171
Title: Development of Precision Nutrition Counseling in Type 2 Diabetes Patients: Using Continuous Glucose Monitoring System
Brief Title: Precision Nutrition Counseling in Type 2 Diabetes Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Seoul National University Hospital (Other)
Collaborators: ChunLab (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: H-1911-059-1078
Record Dates: First submitted 2020-02-02; First posted 2020-02-12 (Actual); Last update posted 2020-02-12 (Actual); Status verified 2020-01

CONDITIONS: Type 2 Diabetes
Keywords: continuous glucose monitor; diet education; Precision nutrition
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CGMS Diet Education (Experimental)
  Interventions: Behavioral: Diet education based on CGMS data
- Conventional Diet Education (Active Comparator)
  Interventions: Behavioral: Conventional diet education

INTERVENTIONS:
Behavioral: Diet education based on CGMS data — Intervention group will receive diet education based on CGMS data, using post prandial glucose response, calculated by incremental area under curve of glucose level. Control group will receive conventional diabetes diet education without CGMS data.
  Arms: CGMS Diet Education
Behavioral: Conventional diet education — Control group will receive conventional diabetes diet education without CGMS data.
  Arms: Conventional Diet Education

SUMMARY:
The aim of this study is to evaluate the effect of precision nutrition education using continuous glucose monitoring system (CGMS) in longterm glycemic control in patients with type 2 diabetes mellitus. Glucose levels in subjects who received diet education using CGMS will be compared to those in subjects who received conventional diet education.

DETAILED DESCRIPTION:
Fifty subjects with type 2 diabetes will be recruited. Every subject will be randomized in two groups, which are CGMS education group and conventional education group. The study will be conducted for 12 weeks for each participants. Intervention group will receive diet education based on CGMS data, using post prandial glucose response, calculated by incremental area under curve of glucose level. Control group will receive conventional diabetes diet education without CGMS data. Primary outcome is change of HbA1c from baseline for 12 weeks, and secondary outcomes are changes of fasting blood glucose level, body weight, waist circumference, blood lipid level, homeostatic model assessment of insulin resistance (HOMA-IR) , c-peptide, microbiome, 7-point self monitoring of blood glucose (SMBG), and compliance/satisfaction questionnaire from baseline for 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes patients (Fasting blood glucose ≥ 126 mg/dl or HbA1c ≥ 6.5% or Subjects who were previously diagnosed with type 2 diabetes and who have been treated with lifestyle modification only, oral anti-diabetic drugs or basal insulin)
* HbA1c 6.5%~10%
* Body weight change less than 5% in 3 month
* Subjects who agreed to the study protocol

Exclusion Criteria:

* Type 1 diabetes patients
* Subjects using insulin other than basal insulin
* Subjects who have newly started or have changed anti diabetic drugs within 3 months
* Subjects who have been received diabetes diet education within 6 months
* Females who are pregnant or doing breast feeding
* Subjects with alcohol addiction or drug abuse
* Subjects who are using drugs that can influence blood glucose levels (e.g. steroid)
* Subjects who are currently using acetaminophen or who should use acetaminophen during CGMS attach period
* Subjects who have skin problems on CGMS sensor insertion site (e.g. burn, excessive body hair, inflammation, rash, tattoo)
* Subjects who have newly started, changed, or stoped probiotics or prebiotics within 2 weeks
* Subjects who have used antibiotics (oral or intravenous) within 2 weeks
* In addition, if it falls under the exclusion criteria according to researchers discretion

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2020-01-16 (Actual); Primary Completion 2021-12-31 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in HbA1c from baseline | 0 week, 12 weeks

SECONDARY OUTCOMES:
Change in fasting blood glucose level from baseline | 0 week, 12 weeks
Change in body weight from baseline | 0 week, 12 weeks
Change in waist circumference from baseline | 0 week, 12 weeks
Change in blood Triglyceride level from baseline | 0 week, 12 weeks
Change in blood High-density lipoprotein level from baseline | 0 week, 12 weeks
Change in blood Low-density lipoprotein level from baseline | 0 week, 12 weeks
Change in HOMA-IR from baseline | 0 week, 12 weeks
Change in c-peptide from baseline | 0 week, 12 weeks
Change in microbiome profile from baseline | 0 week, 12 weeks
  Change in the diversity index of the gut microbiota, change in the compositions of the gut microbiota
Change in 7-point SMBG from baseline | 0 week, 12 weeks
Compliance/Satisfaction Questionnaire | 0 week, 12 weeks
  Change in dietary habits, self-efficacy of diet management , and satisfaction with the education

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No